CLINICAL TRIAL: NCT06646536
Title: The Effect of Anti-Gravity Treadmill Training on Symptoms and Functions in Patients With Meniscus Tears
Brief Title: The Effect of Anti-Gravity Treadmill Training in Patients With Meniscus Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Kübra Alpay, Lecturer of Physiotherapy and Rehabilitation Department, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA24-4
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Meniscus Tear
Keywords: meniscus; anti-gravity; exercise
MeSH Terms: conditions — Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anti-gravity Treadmill Group (Experimental): Anti-gravity treadmill (Alter G) walking program in addition to physiotherapy and rehabilitation
  Interventions: Other: Anti-gravity treadmill training; Other: Standard physiotherapy and rehabilitation program
- Conventional Treadmill Group (Active Comparator): Standard treadmill walking program in addition to physiotherapy and rehabilitation
  Interventions: Other: Conventional treadmill training; Other: Standard physiotherapy and rehabilitation program
- Control Group (Active Comparator): Physiotherapy and rehabilitation program
  Interventions: Other: Standard physiotherapy and rehabilitation program

INTERVENTIONS:
Other: Anti-gravity treadmill training — Patients will participate to anti-gravity treadmill (Alter G) walking program in addition to physiotherapy and rehabilitation program for 6 weeks, 2 days a week.
  Arms: Anti-gravity Treadmill Group
Other: Conventional treadmill training — Patients will participate to walking program on a standard treadmill in addition to physiotherapy and rehabilitation program for 6 weeks, 2 days a week.
  Arms: Conventional Treadmill Group
Other: Standard physiotherapy and rehabilitation program — Patients will participate to physiotherapy and rehabilitation program for 6 weeks, 2 days a week.

SUMMARY:
The aim of this study is to evaluate the effect of anti-gravity treadmill training on symptoms and functions in patients with meniscus tears.

DETAILED DESCRIPTION:
Meniscus tears are one of the most common sports-related injuries. Acute trauma-related tears are more common in active young individuals and athletes. Symptoms such as pain, effusion, tenderness at the joint line, locking, and knee dysfunction are observed after injury. It is aimed to provide painless movement, normal knee kinematics, and retaining of muscle strength in rehabilitation process. Anti-gravity treadmills use an inflatable space around the lower extremities and significantly reduce body weight during walking and running. Anti-gravity treadmill training protects the joint and surrounding soft tissues against the negative effects of loading during the post-injury recovery process, and allows the tissues to heal safely. The aim of this study is to evaluate the effect of anti-gravity treadmill training on symptoms and functions in patients with meniscus tears.

Patients will be randomly divided into three groups: Anti-Gravity Treadmill Group, Conventional Treadmill Group, and Control Group. All patients will be included physiotherapy and rehabilitation program for 6 weeks, 2 days a week. While subjects in the Anti-Gravity Treadmill Group will participate to training anti-gravity treadmill walking, subjects in the Conventional Treadmill Group will participate walking program on a standard treadmill. Symptoms and functions will be assessed baseline and after 6-week program.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years old
* Clinical history and symptoms consistent with MRI-confirmed meniscus tear

Exclusion Criteria:

* History of previous knee surgery
* Other knee ligament pathologies
* Neurological disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale-pain | Baseline, 6 weeks
  Patients will be asked to mark the intensity of the pain they feel on a 10 cm line, where "0" means no pain and "10" means very severe pain.
Knee Injury and Osteoarthritis Outcome Score | Baseline, 6 weeks
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is used to assess symptoms and functional status in knee injuries and osteoarthritis and consists of five dimensions. Each dimension is scored separately and transformed to a scale from 0 to 100. Lower scores from the scale indicate worse pain, symptoms, function, and quality of life.
Dynamic stability | Baseline, 6 weeks
  The single leg dynamic stability will be assessed by using Biodex Balance System® (Biodex Medical Systems, Inc. USA). Low values of the stability index indicate better balance and stability.
Single leg-hop test | Baseline, 6 weeks
  In the single-leg hop test, the measurement of the landing distance from the starting line is recorded for evaluation.

SECONDARY OUTCOMES:
Western Ontario Meniscal Evaluation Tool | Baseline, 6 weeks
  The Western Ontario Meniscal Evaluation Tool (WOMET) is a disease-specific assessment tool used to assess health-related quality of life in patients with meniscus pathology. The least symptomatic score is 0, and the most symptomatic score possible is 1,600. Higher scores indicate a more symptomatic condition.
Kinesiophobia | Baseline, 6 weeks
  The Tampa Kinesiophobia Scale will be used to evaluate kinesiophobia. Scores obtained from the scale range from 17 to 68, with higher scores indicating greater severity of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Alpay, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Eyup, Turkey (Türkiye)